CLINICAL TRIAL: NCT03841305
Title: Simultaneous Portal and Hepatic Vein Embolization Versus Portal Vein Embolization for Hypertrophy of the Future Liver Remnant Before Major Hepatectomy of Non-cirrhotic Liver : a Multicentric Comparative Randomized Phase II Trial
Brief Title: Simultaneous Portal and Hepatic Vein Versus Portal Vein Embolizations for Hypertrophy of the Future Liver Remnant
Acronym: HYPER-LIV01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL18_0025; UF 7595 (Other: UH Montpellier)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: Liver; Interventional radiology; Portal vein embolization; Portal and hepatic vein embolization; Future liver remnant; Surgery; Non-cirrhotic liver; Liver metastases; Colorectal cancer; Liver Regeneration; Liver resection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- portal vein embolization (Active Comparator): Liver preparation before major hepatectomy : portal vein embolization (PVE) in patient with liver metastases from colo-rectal origin considered as resectable.
  Interventions: Procedure: Liver preparation before major hepatectomy
- liver venous deprivation (Experimental): Liver preparation before major hepatectomy : Patients with the liver venous deprivation (LVD) technique that combines both PVE and hepatic vein embolization (HVE) during the same procedure.
  Interventions: Procedure: Liver preparation before major hepatectomy

INTERVENTIONS:
Procedure: Liver preparation before major hepatectomy — Simultaneous portal and hepatic vein embolization versus Portal vein embolization, also called venous deprivation OR portal vein embolization.

SUMMARY:
The hypothesis is that liver venous deprivation (LVD) could strongly improve hypertrophy of the future remnant liver (FRL) at 3 weeks, as compared to portal vein embolization (PVE) in patient with liver metastases from colo-rectal origin considered as resectable.

DETAILED DESCRIPTION:
Portal vein embolization (PVE) has been widely used to generate hypertrophy of the nonembolized lobe in patients undergoing major hepatectomy in order to prevent small-for-size remnant liver resulting in post-operative liver insufficiency.

Although PVE is a safe and effective procedure, it does not always induce sufficient hypertrophy of the future remnant liver (FRL) even after a long time. In case of insufficient liver regeneration following PVE, some authors suggested to embolize hepatic vein(s) (Hwang, Ann Surg 2009).

Interestingly, the sequential right hepatic vein embolization (HVE) after right PVE demonstrated an incremental effect on the FRL. Although attractive, this approach requires two different procedures and does not spare time as compared to PVE alone.

To shorten and optimize the phase of liver preparation before surgery,the so-called liver venous deprivation (LVD) technique that combines both PVE and HVE during the same procedure was developed.

The aim of this randomized phase II trial is to compare the percentage of change in FRL volume at 3 weeks after LVD or PVE using MRI or CT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Liver metastases from colo-rectal origin considered as resectable (as validated by a multidisciplinary committee with at least one senior hepatic surgeon) provided sufficient FRL volume
* Percentage of FRL volume < 30%
* Age ≥ 18 years
* General health status World Health Organisation 0,1
* Estimated life expectancy > 3 months
* Patients whose biological parameters are :

  * Platelets ≥100,000/mm3,
  * Polynuclear neutrophils ≥ 1000/mm3,
  * Hemoglobin≥ 9g/dL (even transfused patients can be included)
  * Creatininemia < 1.5 times the normal value
  * Creatinine clearance > 30 milliliters (mL)/min
  * Bilirubinemia ≤ 1,5 times the normal value
  * liver transaminases ≤ 5 times the normal value
  * prothrombin rate > 70%
* Reference liver CT-Scan or MRI done during the 30 days preceding PVE or LVD.
* Written informed consent
* National health insurance cover

Exclusion criteria

* Patient with cirrhosis
* Presence of clinical ascites
* Ongoing participation or participation within the 21 days prior to inclusion in the study in another therapeutic trial with an experimental drug
* Serious non-stabilized disease, active uncontrolled infection or other serious underlying disorder likely to prevent the patient from receiving the treatment
* Pregnancy (betaHCG positive), breast-feeding or the absence of effective contraception for women of child-bearing age
* Contraindication for the MRI : Pacemaker or neurosensorial stimulator or implantable defibrillator, cochlear implant, ferromagnetic foreign body similar to the nervous structure.
* Allergy or contra-indication to iodine contrast agents (thyrotoxicosis, allergy to the active substance or excipients)
* Treatment with anticoagulants (heparin or AVK) that cannot be interrupted for 48 hours
* Treatment with anti-platelets that cannot be interrupted for 5 days for aspirin or Plavix
* Legal incapacity (persons in custody or under guardianship)
* Deprived of liberty Subject (by judicial or administrative decision)
* Impossibility to sign the informed consent document or to adhere to the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
increase in volume of the future remnant liver (FRL) | at 3 weeks after liver venous deprivation (LVD) or portal vein embolization (PVE) using MRI or CT-scan
  The primary outcomes is to compare the increase in volume of the future remnant liver (FRL)

SECONDARY OUTCOMES:
Tolerance | between the day of liver preparation and 90 days after surgery
  Toxicities are evaluated according to NCI-CTCAE version 4.03 published 14 June 2010
Post-operative mortality | 90 days after surgery
  Post-operative mortality defined as any death within 90 days after surgery or within the hospital stay
Post-operative morbidity | 90 days after surgery
  Post-operative morbidity defined as the percentages of grade I/II/III/IV/V complications according to Clavien-Dindo classification within the 90 days after surgery or within the hospital stay.
Post-hepatectomy liver failure | between the day of the surgery and 90 days after surgery
  Post-hepatectomy liver failure defined according to the "50-50" criteria or peak bilirubin >7mg/dL.
Rate of non-resectability due to insufficient FRL | between the day of the treatment and the day of the surgery
  Rate of non-resectability due to insufficient FRL defined as the percentage of patients for whom resection will be not attempted due to insufficient FRL
Rate of non-resectability due to tumor progression | between the day of the treatment and the day of the surgery
  Rate of non-resectability due to tumor progression defined as the percentage of patients for whom resection will not be attempted due to tumor progression.
Rate of per-operative difficulties | between the day of the surgery and 90 days after surgery
  Rate of per-operative difficulties defined as the percentage of patients for whom per-operative difficulties are encountered by the surgeon
Blood loos, operating time, transfusion | the day of the surgery
  Blood loss are evaluated in mL. Operating time avec evaluated in minutes and transfusion are evaluated by number of packed red blood cells
R0 resection rate | the day of the surgery
  Rate of R0 resection defined as no microscopic tumor residual
R1 resection rate | the day of the surgery
  Rate of R1 resection defined as the percentage of patients resected with margin <1mm
Pre and post-operative liver volumes | Baseline, week 1, week 3 then every 2 weeks until surgery or week 7 and 4 weeks after surgery
  Pre and post-operative liver volumes will be evaluated through CT or MRI acquisitions by calculating whole liver, tumor and FRL volumes
Recurrence-free survival | 90 days after surgery
  Recurrence-free survival defined as the time from date of randomization to date of recurrence or death from their tumor. Patients alive will be censored at the date of last news.
Overall survival | Between the liver preparation and 90 days after surgery
  Overall survival defined as the time from date of randomization to date of death from any cause. Patients alive will be censored at the date of last news.
Evaluation of pre and post-operative liver function | Baseline, week 1, week 3 then every 2 weeks until surgery or week 7 and 4 weeks after surgery
  Evaluation of pre and post-operative liver function will be evaluated using 99mTc mebrofenine scintigraphy through SPECT/CT acquisitions by calculating mebrofenin clearance in %/min/m² of whole liver and FRL at the same time points as CT/MRI
To search for biomarkers predictive of liver hypertrophy/regeneration and immune cell response | The day of liver preparation, on day 1, day 2 and day 3 after liver preparation and the day of surgery
  Biomarkers predictive of liver hypertrophy/regeneration are evaluated by blood samples and liver biopies

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Montpellier, Montpellier, Hérault
  - CHU d'Angers, Angers
  - Bordeaux University Hospital, Bordeaux
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Centre Léon Berard, Lyon
  - CHU de Nice, Nice
  - APHP - Cochin hospital, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Deshayes E, Piron L, Bouvier A, Lapuyade B, Lermite E, Vervueren L, Laurent C, Pinaquy JB, Chevallier P, Dohan A, Rode A, Sengel C, Guillot C, Quenet F, Guiu B. Study protocol of the HYPER-LIV01 trial: a multicenter phase II, prospective and randomized study comparing simultaneous portal and hepatic vein embolization to portal vein embolization for hypertrophy of the future liver remnant before major hepatectomy for colo-rectal liver metastases. BMC Cancer. 2020 Jun 19;20(1):574. doi: 10.1186/s12885-020-07065-z. PMID 32560632